CLINICAL TRIAL: NCT05876897
Title: Correlation Between MRI and Ultrasound for Diagnosis of Lower Limb Bone Stress Injuries
Brief Title: US vs MRI for Stress Injuries
Status: Completed | Type: Observational
Sponsor: Ryan Kruse (Other)
Responsible Party: Sponsor-Investigator, Ryan Kruse, Clinical Assistant Professor, University of Iowa
Organization: University of Iowa (Other)
Other Study IDs: 202010068
Record Dates: First submitted 2023-05-14; First posted 2023-05-26 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Stress Fracture
MeSH Terms: conditions — Fractures, Stress

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Diagnostic Ultrasound

SUMMARY:
The primary purpose of this study is to determine whether or not there is a correlation between MRI and ultrasound for the diagnosis of lower limb stress injuries. Patients that are seen at the University of Iowa Sports Medicine Center with a suspected diagnosis of a lower limb stress injury will be recruited. These patients will undergo a diagnostic ultrasound of the affected region prior to undergoing an MRI of that region. Then, the ultrasound findings will be compared to the MRI findings to determine if a correlation exists.

ELIGIBILITY:
Inclusion criteria:

* Age 18-50
* MRI confirmed tibial or metatarsal stress injury

Exclusion criteria:

-Prior history of stress fracture or fracture in the affected limb at the region of concern.

Ages: 18 Years to 50 Years | Sex: All
Age Groups: Adult
Study Population: 25 patients ages 18-50 with a suspected diagnosis of a lower limb stress injury (specifically of the tibia or metatarsal) will be recruited. Patients will excluded if they have a prior history of stress fracture or fracture in the affected limb at the region on concern.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2021-02-03 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
US correlation to MRI | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- University of Iowa Sports Medicine, Iowa City, Iowa, United States